CLINICAL TRIAL: NCT07091643
Title: Neuroimaging Markers of Midlife Depression and Cognitive Behavioural Therapy (CBT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Jean Chen, Senior Scientist, Baycrest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB 22-10
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Midlife Depression; Depression; Cognitive Behavioural Therapy (CBT)
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Individuals with midlife depression (MDD, ages 40-60 years) will undergo 12 weeks of CBT, in addition to three follow-up assessments, clinical evaluation (including completion of self-report and clinician-rated questionnaires) and pre-post CBT magnetic resonance imaging (MRI).
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — 12 weeks of Cognitive Behavioural Therapy (CBT) will be administered. The first session will be accomplished in-person at Baycrest Hospital. After that, therapy will be conducted virtually, via video-conference. Individuals will undergo therapy once a week for approximately 1 hour, for 12-weeks. Following the 12-week period, individuals will receive three follow-up assessments with their therapist at 3, 6, and 9 months.

SUMMARY:
Major depressive disorder (MDD) is associated with significant cognitive impairment throughout the life-course, which may progress toward MCI and dementia with age. Antidepressant medications are the first line of treatment; however, they fail to adequately address cognitive deficits and prevent relapse. Sustained cognitive impairment into euthymic periods may relate to underlying neurobiological changes, which could potentially be addressed through Cognitive Behavioural Therapy (CBT). Notably, CBT has been shown to improve cognitive domains including divided attention, memory, and processing speed while preventing depression relapse. Midlife represents a critical period in which shared neurobiological factors (such as brain changes on a vascular, morphological, and functional level) underlying depression and cognitive impairment could accelerate toward MCI and dementia. An updated understanding of neurobiological correlates of midlife depression and CBT response through multimodal neuroimaging is critical to improving affective and cognitive outcomes in this population.

The overarching objective of this project is to use multimodal neuroimaging to quantify the neurobiological and clinical impact of CBT in midlife depression. Specifically, we aim to:

1. Investigate the clinical impact of CBT on cognitive function and mood outcomes in midlife depression
2. Examine functional connectivity and microstructural determinants of CBT response in midlife depression using neuroimaging
3. Identify vascular modulators of neural connectivity and CBT response in midlife depression.

We hypothesize that midlife depression will be associated with functional and structural neural connectivity changes, which will be accompanied by vascular pathology. Adequate CBT response (i.e., improvements in mood and cognitive function) will be associated with amelioration of neurobiological changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-60 years, inclusive.
2. Diagnosis of MDD as per the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)6 determined through a structured clinical interview.
3. Current major depressive episode of at least 3 months in length.
4. Depression of at least mild severity defined by a total score of ≥7 on the Montgomery Asberg Depression Rating Scale (MADRS)7.
5. Ability to understand and comply with the requirements of the study, as judged by the investigator(s).

Exclusion Criteria:

1. Presence of comorbid post-traumatic stress disorder, obsessive-compulsive disorder, eating disorder(s), schizophrenia, or other psychiatric disorders.
2. History of a manic, hypomanic, or mixed depressive episode.
3. Treatment with electroconvulsive therapy, intravenous and/or intranasal ketamine in the 6-weeks prior to study enrolment.
4. History of substance-use disorder in the past 12 months.
5. Presence of current alcohol-use disorder
6. A positive urine toxicology screen for non-prescribed substance use.
7. A positive pregnancy test at screening.
8. A history of major medical or neurological illness.
9. A history of traumatic brain injury, stroke, seizures, or previous brain surgery.
10. Contraindications to magnetic resonance imaging (MRI) scanning.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MADRS | Once before administration of Cognitive Behavioural Therapy (CBT) and once after (baseline and 12 weeks).
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated scale used to assess the severity of depressive symptoms. It is a 10-item scale, with each item rated on a 7-point scale, and the total score ranges from 0 to 60, with higher scores indicating more severe depression. The MADRS is commonly used in clinical trials and research to evaluate treatment response in individuals with depression.
DARS | Once before administration of Cognitive Behavioural Therapy (CBT) and once after (baseline and 12 weeks).
  The Dimensional Anhedonia Rating Scale (DARS) is a 17-item self-report scale used to assess anhedonia, a core symptom of depression characterized by a reduced ability to experience pleasure. It measures anhedonia across four domains: hobbies, food/drink, social activities, and sensory experiences, evaluating aspects like desire, motivation, effort, and consummatory pleasure.

SECONDARY OUTCOMES:
T1-anatomical | Once before administration of Cognitive Behavioural Therapy (CBT) and once after (baseline and 12 weeks).
  A T1 anatomical MRI, also known as a T1-weighted MRI, is a type of magnetic resonance imaging (MRI) sequence that excels at visualizing the structural details of tissues, particularly soft tissues and fat. It's often used to provide a clear view of the b
Diffusion-tensor MRI | Once before administration of Cognitive Behavioural Therapy (CBT) and once after (baseline and 12 weeks).
  Diffusion tensor MRI (DTI) is an advanced magnetic resonance imaging (MRI) technique that maps the diffusion of water molecules in the brain to visualize the white matter pathways. It provides insights into the structural organization and integrity of white matter, which is crucial for understanding brain connectivity and function.
Resting-state fMRI | Once before administration of Cognitive Behavioural Therapy (CBT) and once after (baseline and 12 weeks).
  Resting state fMRI (rs-fMRI) is a technique used to study brain activity when a person is not performing a specific task. It focuses on spontaneous fluctuations in the blood-oxygen-level-dependent (BOLD) signal to identify functional connections between different brain regions. We will use this signal to compute functional connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- Baycrest Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] World Health Organization. Division of Mental Health and Prevention of Substance Abuse. (1997). WHOQOL : measuring quality of life. World Health Organization.
- [Background] Leach, L., Kaplan, E., Rewilak, D., Richards, B., & Proulx, G. (2000). The Kaplan-Baycrest neurocognitive assessment (KBNA): Test manual. San Antonio, TX, Harcourt Assessment.
- [Background] Soares CN. Mood disorders in midlife women: understanding the critical window and its clinical implications. Menopause. 2014 Feb;21(2):198-206. doi: 10.1097/GME.0000000000000193. PMID 24448106
- [Background] Perini G, Cotta Ramusino M, Sinforiani E, Bernini S, Petrachi R, Costa A. Cognitive impairment in depression: recent advances and novel treatments. Neuropsychiatr Dis Treat. 2019 May 10;15:1249-1258. doi: 10.2147/NDT.S199746. eCollection 2019. PMID 31190831
- [Background] Brenowitz WD, Zeki Al Hazzouri A, Vittinghoff E, Golden SH, Fitzpatrick AL, Yaffe K. Depressive Symptoms Imputed Across the Life Course Are Associated with Cognitive Impairment and Cognitive Decline. J Alzheimers Dis. 2021;83(3):1379-1389. doi: 10.3233/JAD-210588. PMID 34420969